CLINICAL TRIAL: NCT03635905
Title: Gabapentin as an Adjunct for Pain Management During Dilation and Evacuation: A Double-blind Randomized Controlled Trial
Brief Title: Gabapentin for Pain Management During Dilation and Evacuation
Acronym: Gabapentin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Society of Family Planning Research Fund (Unknown)
Responsible Party: Principal Investigator, Pamela Lotke, Principal Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-092
Record Dates: First submitted 2018-07-20; First posted 2018-08-17 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Pain
Keywords: abortion; gabapentin; Neurontin; Dilation and evacuation
MeSH Terms: conditions — Pain; Dilatation, Pathologic | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin (Neurontin)- 600 mg oral administered pre-operatively at the time of cervical preparation
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin (Neurontin®) is FDA-approved for the treatment of post-herpetic neuralgia and seizure disorder. Off-label uses include chronic refractory cough, neuropathy, hot flashes, restless leg syndrome, social anxiety disorder, and post-operative pain
  Other Names: (Neurontin)
  Arms: Gabapentin
Drug: Placebo — Methylcellulose placebo capsule
  Arms: Placebo

SUMMARY:
Justification. Pain control is still an issue for women undergoing second trimester abortion procedures. The investigators propose a randomized controlled double-blinded trial evaluating the use of adjunct gabapentin versus placebo in addition to moderate sedation during D&E. The investigators hypothesize that 600 mg oral gabapentin administered pre-operatively at the time of cervical preparation initiation will improve intra-operative pain control. The investigators also hypothesize that it will improve pre- and post-operative pain, anxiety, nausea, vomiting, and overall satisfaction with pain management during D&E.

To test the hypotheses the investigators plan to enroll 130 participants who will be randomized 1 to 1 to receive either 600 mg gabapentin or placebo at the initiation of cervical preparation.

DETAILED DESCRIPTION:
Over 900,000 abortion procedures are performed annually in the United States [1]. For many women, pain relief during abortion is inadequate despite the use of non-steroidal anti-inflammatory drugs, local anesthetics, opioids, and/or moderate sedation. Research on pain control during abortion has focused on methods for relief during first-trimester suction curettage with little research dedicated to pain during dilation and evacuation (D&E). Gabapentin (Neurontin) has emerged as an effective adjunct to pain management for a variety of surgical procedures. Gabapentin is inexpensive and is also effective in reducing anxiety, nausea, and vomiting. The addition of pre-operative gabapentin to moderate sedation during D&E may lead to increased patient satisfaction and pain relief without significantly increasing risk or cost.

Proposed Research. The investigators propose a randomized controlled double-blinded trial evaluating the use of adjunct gabapentin versus placebo in addition to moderate sedation during D&E. The investigators hypothesize that 600 mg oral gabapentin administered pre-operatively at the time of cervical preparation initiation will improve intra-operative pain control. The investigators also hypothesize that it will improve pre- and post-operative pain, anxiety, nausea, vomiting, and overall satisfaction with pain management during D&E. The investigators hypothesize that the doses of moderate sedation agents required to obtain adequate sedation will be decreased if participants receive gabapentin, versus placebo. The investigators also plan to compare the risk of adverse events with adjunct gabapentin versus placebo with moderate sedation.

To test the hypotheses the investigators plan to enroll 130 participants who will be randomized 1 to 1 to receive either 600 mg gabapentin or placebo at the initiation of cervical preparation. Baseline characteristics will be recorded. Pain will be assessed pre-operatively, at 3 intraoperative time points, and postoperatively by 100 mm visual analog scale (VAS). The investigators plan to assess satisfaction with pain control, nausea, vomiting, and anxiety preoperatively and post-operatively, using 5-point Likert scales and the State Trait Anxiety Inventory, respectively. A final assessment will be made by phone on post-operative day one to evaluate overall satisfaction and perform a final screen for adverse events.

New features. No publications have evaluated the use of gabapentin during abortion care, although multiple studies are currently underway investigating gabapentin's effects during first trimester abortion and during overnight cervical osmotic dilators. To the investigators knowledge, this will be the first evaluation of gabapentin in conjunction with moderate sedation for pain relief during same-day second trimester abortion.

ELIGIBILITY:
Inclusion Criteria:

* English proficiency
* 18 years of age or older
* Gestational age 14 weeks or greater
* Ability to provide informed consent
* Desire to proceed with outpatient D&E under moderate sedation

Exclusion Criteria:

* Contraindications to outpatient abortion or moderate sedation
* Current use of gabapentin (Neurontin®) or pregabalin (Lyrica®)
* Severe renal disease
* Allergy or sensitivity to gabapentin or pregabalin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Maximum procedural pain | Intra-operative
  Measured on 100-mm visual analog scale (higher score = more pain)

SECONDARY OUTCOMES:
Peri-operative pain | At enrollment, prior to procedure, speculum insertion, aspiration, speculum removal, and discharge from clinic, usually within 30 to 120 minutes after completion of procedure.
  Measured by 100-mm visual analog scale (higher score represents more pain)
Nausea | At enrollment, prior to procedure, speculum insertion, aspiration, speculum removal, and discharge from clinic, usually within 30 to 120 minutes after completion of procedure.
  Measured on 5-point Likert scale (higher score represents more nausea)
Vomiting | At enrollment, prior to procedure, speculum insertion, aspiration, speculum removal, and discharge from clinic, usually within 30 to 120 minutes after completion of procedure.
  Measured on 5-point Likert scale (higher score represents more vomiting)
Anxiety | Prior to procedure and prior to discharge from clinic, usually within 30 to 120 minutes after completion of procedure.
  Measured by State Trait Anxiety Inventory. 20 State anxiety items. Higher score represents more anxiety
Satisfaction with pain management | Prior to procedure, prior to discharge from clinic, usually within 30 to 120 minutes after completion of procedure, and post-operative day 1
  Measured on 5-point Likert scale (Higher score represents greater satisfaction)
Adverse events | Recorded on day of procedure and post-operative day 1
  Including but not limited to respiratory depression and sedation reversal
IV sedation doses | Day of procedure
  Doses of IV fentanyl and IV midazolam administered

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Planned Parenthood, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brant AR, Reeves MF, Ye PP, Scott RK, Floyd S, Tefera E, Lotke PS. Gabapentin as an adjunct for pain management during dilation and evacuation: A double-blind randomized controlled trial. Contraception. 2023 Feb;118:109892. doi: 10.1016/j.contraception.2022.09.130. Epub 2022 Oct 12. PMID 36243129